CLINICAL TRIAL: NCT00136734
Title: Methylphenidate Treatment for Cocaine Abuse and ADHD
Brief Title: Methylphenidate Treatment for Cocaine Abuse and ADHD - 1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Frances R Levin, Director of Substance Use Disorder, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: #3236-NIDA-011755-1; R01DA011755 (NIH)
Record Dates: First submitted 2005-08-25; First posted 2005-08-29 (Estimated); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Attention Deficit Disorder With Hyperactivity; Cocaine-Related Disorders
Keywords: ADHD; Cocaine dependence; treatment; methylphenidate
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Cocaine-Related Disorders | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): methylphenidate
  Interventions: Drug: Methylphenidate
- 2 (Placebo Comparator): placebo
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Methylphenidate
  Arms: 1
Other: placebo — placebo
  Arms: 2

SUMMARY:
Many cocaine dependent individuals are also diagnosed with Attention Deficit Hyperactivity Disorder (ADHD). Methylphenidate (Ritalin) is currently approved to treat individuals diagnosed with ADHD. The purpose of this study is to determine the effectiveness of methylphenidate in treating ADHD symptoms in cocaine dependent individuals.

DETAILED DESCRIPTION:
Methylphenidate (MPH) is commonly used to treat individuals diagnosed with ADHD. The purpose of this study is to determine the effectiveness of MPH in treating adult cocaine dependent individuals who are also diagnosed with ADHD.

Participants in this 14-week, double-blind, placebo-controlled study will be randomly assigned to receive either sustained-release MPH or placebo. All participants will receive individual cognitive behavioral therapy. The trial will last 14 weeks. It will include a 1-week placebo lead-in phase and a 2-week dose titration phase, followed by 11 weeks on a stable dose of MPH. During the titration phase, MPH will be given twice a day, starting at a dose of 10 mg/day. The dose will increase by 10 mg each day, until a final stable dose of 40 mg/day is reached. At this time, sustained-release MPH will be given as two 20 mg doses (one in the morning and one in the afternoon). Depending on a participant's tolerance of MPH, the dose will be increased to a maximum of 60 mg/day (40 mg in the morning and 20 mg in the afternoon). Participants who are unable to tolerate a dose of at least 40 mg/day of MPH will be discontinued from the study. Assessments of ADHD symptoms will be completed at weekly study visits. In addition, drug use assessments will also be completed and will include self-reports and urine toxicology tests.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for cocaine dependence
* Meets DSM-IV criteria for persistent adult Attention Deficit Hyperactive Disorder

Exclusion Criteria:

* Meets DSM-IV criteria for current psychiatric disorders (other than ADHD or substance abuse) that requires a psychiatric intervention
* Physiologically dependent on sedatives or alcohol, to the extent that medical attention is required during periods of abstinence or significant reduction in the amount of use
* Exhibits suicidal or homicidal behavior within the two years prior to enrollment
* Currently taking prescription psychotropic medication
* Unstable medical condition (e.g., uncontrolled diabetes) that would make participation in the study hazardous
* Known sensitivity to methylphenidate
* Pregnant or breastfeeding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 124 (Actual)
Dates: Start 1998-04; Primary Completion 2004-03 (Actual); Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
ADHD symptom severity based on the ADHD rating scale score | measured weekly for the 14 weeks of the trial or length of study participation
self reported cocaine use | recorded daily for the 14 weeks of the trial or the length of participation

CONTACTS AND LOCATIONS:
Overall Officials: Frances R Levin, M.D., Principal Investigator — Research Foundation for Mental Hygiene, Inc.
Locations (1):
- Research Foundation for Mental Hygiene, Inc., New York, New York, United States

REFERENCES:
- [Result] Levin FR, Evans SM, Brooks DJ, Garawi F. Treatment of cocaine dependent treatment seekers with adult ADHD: double-blind comparison of methylphenidate and placebo. Drug Alcohol Depend. 2007 Feb 23;87(1):20-9. doi: 10.1016/j.drugalcdep.2006.07.004. Epub 2006 Aug 22. PMID 16930863
- See also: Related Info — http://stars.columbia.edu